CLINICAL TRIAL: NCT00837668
Title: Stromal Gene Expression During Pulmonary Sarcoidosis
Status: Terminated | Type: Observational
Why Stopped: Interim analysis
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Elliott Crouser MD, Associate Professor of Internal Medicine, Ohio State University
Other Study IDs: 2005H0018
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Sarcoidosis
Keywords: sarcoidosis; stromal gene expression; pulmonary sarcoidosis; bronchoscopy
MeSH Terms: conditions — Sarcoidosis; Sarcoidosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sarcoidosis: sarcoidosis patients undergoing clinical bronchoscopy

SUMMARY:
to determine the genetic pathways operating at the tissue level to cause granulomatous inflammation in the lungs and lymph nodes of patients with sarcoidosis. By so doing, we hope to identify unique genetic mechanisms which will aid in the diagnosis of sarcoidosis and will help us understand the pathogenesis of this poorly understood disease.

DETAILED DESCRIPTION:
to collect small sample of lung tissue recovered from a clinical procedure such as bronchoscopy, or a mediastinoscopy (a procedure in which a lighted instrument (mediastinoscope) is inserted through a neck incision to visually examine the structures in the top of the chest cavity and to take a sample (biopsy) of tissue.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sarcoidosis

Exclusion Criteria:

* inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from sarcoidosis clinic
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2005-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To Identify Gene Expression Patterns That Specifically Correlate With Active Pulmonary Sarcoidosis. | end of study

SECONDARY OUTCOMES:
To Determine if Gene Expression Patterns Correlate With The Severity of Illness Of Sarcoidosis Patients | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Crouser, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States